CLINICAL TRIAL: NCT05212428
Title: MAYO CLINIC TAPESTRY: Use of Genomic Sequencing in Clinical Practice
Brief Title: DNA Sequencing in Clinical Practice, Mayo Clinic Health Tapestry Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19-000001; NCI-2021-00497 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); TAPESTRY (Other: Study Team)
Record Dates: First submitted 2021-02-04; First posted 2022-01-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Genetic Disorder
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Specimen Handling; Genetic Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (biospecimen collection, genetic analysis) (Experimental): Participants receive a saliva kit, register with Helix then undergo collection of saliva sample which is returned o Helix. Participants also receive an online link to complete the About Me family history. Once sequencing is completed by Helix, ancestry/trait information and genetic findings are shared with participants and their primary provider, if applicable. Participants with positive results are offered genetic counseling and are encouraged to seek clinical confirmatory testing. Following clinical confirmation, results are scanned into the electronic health record. Participants may also undergo the collection of blood, urine, and stool samples for future studies.
  Interventions: Procedure: Biospecimen Collection; Other: Diagnostic Laboratory Biomarker Analysis; Other: Genetic Counseling; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of saliva, blood, urine and stool samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Other: Genetic Counseling — Receive genetic counseling
Other: Questionnaire Administration — Complete family history
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial collects information on how sequencing a patient's deoxyribonucleic acid (DNA) (i.e., the genetic material) could impact their health care. This study also develops and improves ways to include genomic information from DNA sequencing into the electronic health record to create a more complete "Health Tapestry" for each participant. Sequencing of a patient's DNA leads to the detection of genetic variants some of which determine risk for disease development. Discovery of those genetic variants in a patient could result in prevention, earlier diagnosis or better therapy of disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To detect and compare the actionable genetic findings derived from whole exome sequencing (WES) testing and examine their frequency and association with family history using a large cohort of patients seen across specialties within the Mayo Clinic enterprise.

II. To assess the effect of actionable genetic findings of patients on health-care utilization, and patients acceptance.

III. To create a unique vertically integrated data asset (Mayo Clinic Health Tapestry) that links genomics and other omics information to traditional health parameters in the Electronic Medical Record (EMR) with the aim to elucidate disease formation and outcomes.

IV. Assess the frequency of hereditary cancer predisposition genes (BRCA1, BRCA2, Lynch syndrome mismatch repair [MMR] genes) through population screening using WES and the uptake of genetic counseling.

V. To study the genetic predisposition to coronavirus disease 2019 (COVID-19) disease we propose using a COVID-19 survey.

VI. Assess the recruitment rate of those approached by portal and email. VII. Assess differential consent rates by combinations of mode of invitation (initial contact via email or patient portal) and content of material (standard invitation content vs. enhanced content with improved language and visual display) in one cohort.

OUTLINE:

Participants receive a saliva kit, register with Helix then undergo collection of saliva sample which is returned o Helix. Participants also receive an online link to complete the About Me family history. Once sequencing is completed by Helix, ancestry/trait information and genetic findings are shared with participants and their primary provider, if applicable. Participants with positive results are offered genetic counseling and are encouraged to seek clinical confirmatory testing. Following clinical confirmation, results are scanned into the electronic health record. Participants may also undergo the collection of blood, urine, and stool samples for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Registered Mayo Clinic patient
* Able to provide informed written consent
* E-mail and web access (for electronic consent, video education, registering with Helix and receiving results)
* Ability to collect and ship saliva sample within the United States
* Of note: Women, who are pregnant, or planning to become pregnant, can take part in this study. However, this study does not replace prenatal genetic testing. If participants have these concerns, they will be encouraged to contact their obstetrics (OB) provider or a genetic counselor to discuss further

Exclusion Criteria:

* Other co-morbidity which would in physician's opinion interferes with patient's ability to participate in the study (eg: reduced ability to comprehend eg: dementia, intellectual disability, fluency in consent language)
* Allogeneic bone marrow transplant (e.g. samples from autologous bone marrow transplant recipients are acceptable if collected at least one month after transplant)
* Active hematological cancer or history of a hematological cancer
* Resident of the state of New York

  * The Helix lab does not currently have New York state licensure
* Residents without a shipping address in the United States

  * The Helix lab is unable to ship and receive samples internationally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110000 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Actionable genetic findings derived from whole exome sequencing (WES) testing | Up to 5 years
  Patients will be asked to complete a family history as part of this study. The family history will be assessed to determine the percentage of participants with evidence of genetic risk for the actionable finding. Standard descriptive statistics approaches will be used for analysis.
Effect of actionable genetic findings of patients on health-care utilization | Up to 5 years
  Medical records will be reviewed for evidence that patients take active participation in managing genetic risks. Additionally, patients will be surveyed as to their experience with genomic based testing. Standard descriptive statistics approaches will be used for analysis.
Patients' acceptance | Up to 5 years
  Standard descriptive statistics approaches will be used for analysis.
Creation of a unique vertically integrated data asset (Mayo Clinic Health Tapestry) | Up to 5 years
  A variety of patient cohorts will be ascertained throughout this study. Data will be made available to researchers to query correlations of disease states and clinical outcomes to genomic findings. These insights will be invaluable to creating genomic informed care plans in the future. Standard descriptive statistics approaches will be used for analysis.
Genetic predisposition to coronavirus disease 2019 (COVID-19) disease | Up to 5 years
  Will examine the genetic variants derived from the WES data that associate with COVID-19 outcomes. Standard descriptive statistics approaches will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos N. Lazaridis, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Samadder NJ, Schroeder M, Voss MM, Shamoun F, Kullo I, Curry TB, Houwink EJF, Bublitz ML, Bandel LA, Armasu SM, Vierkant RA, Ferber MJ, Olson R, Tan-Arroyo J, Morales-Rosado JA, Klee EW, Larson NB, Kruisselbrink TM, Egan JB, Kemppainen JL, Bidwell JS, Anderson JL, McAllister TM, Baudhuin LM, Kunze KL, Golafshar MA, Presutti RJ, Summer-Bolster JM, Lazaridis KN. Exome Sequencing Enhances Screening for Familial Hypercholesterolemia Within a Multi-Site Healthcare System. Circ Genom Precis Med. 2025 Dec;18(6):e005174. doi: 10.1161/CIRCGEN.125.005174. Epub 2025 Nov 12. PMID 41221644
- [Derived] Bandel LA, Vierkant RA, Kruisselbrink TM, Bublitz ML, Wilson TA, Armasu SM, Egan JB, Presutti RJ, Samadder NJJ, Sekulic A, Olson RJ, Tan-Arroyo J, Morales-Rosado JA, Klee EW, Ferber MJ, Kemppainen JL, Anderson JL, Bidwell JS, Wick JJ, Ortega VE, Bobo WV, Pichurin PN, Mcmillan JM, Weaver DM, Riegert-Johnson DL, Cera AM, Boucher LM, Kullo IJ, Mantia SK, Jones MT, Larson NB, Luehrs TC, Leitzke JW, Sicotte H, Tian S, Stavlund JR, Pacyna JE, Sharp RR, Asabere AA, Lu J, McAllister TM, Walker TS, Stewart AK, Farrugia G, Lazaridis KN. Mayo Clinic Tapestry Study: A Large-Scale Decentralized Whole Exome Sequencing Study for Clinical Practice, Research Discovery, and Genomic Education. Mayo Clin Proc. 2024 Nov 5:S0025-6196(24)00405-1. doi: 10.1016/j.mayocp.2024.08.005. Online ahead of print. PMID 39625429
- [Derived] Samadder NJ, Gay E, Lindpere V, Bublitz ML, Bandel LA, Armasu SM, Vierkant RA, Ferber MJ, Klee EW, Larson NB, Kruisselbrink TM, Egan JB, Kemppainen JL, Bidwell JS, Anderson JL, McAllister TM, Walker TS, Kunze KL, Golafshar MA, Klint MA, Presutti RJ, Bobo WV, Sekulic A, Summer-Bolster JM, Willman CL, Lazaridis KN. Exome Sequencing Identifies Carriers of the Autosomal Dominant Cancer Predisposition Disorders Beyond Current Practice Guideline Recommendations. JCO Precis Oncol. 2024 Jul;8:e2400106. doi: 10.1200/PO.24.00106. PMID 39013133
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials